CLINICAL TRIAL: NCT02283983
Title: Evaluation of Cryoprotection of Nail Toxicity Induced by Docetaxel Low Cumulative Dose. Controlled, Randomized, Open, Multicentre Prospective.
Brief Title: Evaluation of Cryoprotection Induced Nail Toxicity Docetaxel Low Cumulative Dose
Acronym: BANQUISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHD 097-13
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard cryoprotection (Active Comparator): Proposal helmet without mittens and booties
  Interventions: Other: cooling helmet
- Cryoprotection with mittens and booties (Experimental): Standard cryoprotection with mittens and booties
  Interventions: Other: mittens and booties; Other: cooling helmet

INTERVENTIONS:
Other: mittens and booties
  Arms: Cryoprotection with mittens and booties
Other: cooling helmet

SUMMARY:
For the specific patient population studied receiving 5-Fluorouracil, epirubicin and cyclophosphamide - Docetaxel sequence (cumulative dose <300 mg / m2), using a cryoprotection has never been assessed.

The effectiveness of cryoprotection of onycholysis secondary to Docetaxel is not well established in this population (breast cancer in the adjuvant setting) and is based solely on a publication (Scotté) that does not contain the same therapeutic modalities (dose significantly higher). The few studies available have heterogeneous populations, nonrandomized, retrospective or with a small sample.

By extension to what has been observed with higher cumulative doses of docetaxel, some teams offer mittens and booties chilled to their patients, a practice that is not the subject of a national consensus.

The investigators wish to accurately assess the effectiveness of mittens and slippers chilled, their tolerance and their observance because of weak data on this specific population in the literature.

ELIGIBILITY:
Inclusion Criteria:

* upper age to 18 years
* mammary adenocarcinoma nonmetastatic and histologically proven
* wait under an adjuvant or neoadjuvant chemotherapy according to the following conventional scheme: 3 cycles of F5-Fluorouracil, epirubicin and cyclophosphamide 100 (500 or 5-Fluorouracil 600 mg / m² J1, Epirubicin 100 mg / m² J1, Cyclophosphamide 500 or 600 mg / m² J1 or 3 cycles of Epiribucin and Cyclophosphamide 100) followed by 3 cycles of docetaxel, 100 mg / m², +/- trastuzumab if Her2+++
* Patient with the capacity/faculties to understand a newsletter and sign an informed consent
* Patient receiving social coverage
* Patient who can be treated and followed in the center for a period of at least one year
* WHO scale 0 or 1

Exclusion Criteria:

* Age below 18 years
* Diseases of the scalp or whatever hair-showing against helmet or alopecia
* Using pre nail resin before and per chemotherapy
* mammary adenocarcinoma stage IV
* Indication of docetaxel for cancer of another organ than breast
* Treatment processing or programmed during chemotherapy with an innovative molecule being evaluated
* Raynaud's syndrome, cold agglutinin disease, cryoglobulinemia and cryofibrinogenemia.
* Uncontrolled severe arterial disease.
* Presence of a device> grade 1 neuropathy before the start of chemotherapy
* Patient unable to submit the protocol followed for psychological, social, family or geographical
* Patient with an incompatible underlying disease or concomitant with the inclusion in the trial, whether psychiatric or somatic
* Patient trust, guardianship, under legal protection measure, deprived of freedom
* Male
* Criteria for non randomization (before the first course of docetaxel) :

  * Presence of peripheral neuropathy> grade 1 after the first 3 cycles of 5-Fluorouracil, epirubicin and cyclophosphamide 100.
  * Presence of a nail or skin toxicity> grade 1 after 3 cycles of 5-Fluorouracil, epirubicin and cyclophosphamide 100.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank PRIOU, PH, Study Director — CHD Vendee La Roche sur Yon
Locations (10):
- France (10):
  - Institut de cancérologie de l'Ouest - Angers, Angers
  - Centre Hospitalier de Cholet, Cholet
  - CHD Vendee, La Roche-sur-Yon
  - CH du Mans, Le Mans
  - Centre hospitalier Bretagne Sud, Lorient
  - Centre Catherine de Sienne, Nantes
  - Institut de cancérologie de l'Ouest - Nantes, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre d'Oncologie Saint-Yves, Vannes
  - CHBA Vannes, Vannes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 319 enrolled participants, 280 met inclusion criteria and were randomized to treatment
Groups:
- Cryoprotection With Mittens and Booties: Standard cryoprotection with mittens and booties
  mittens and booties
  cooling helmet
- Standard Cryoprotection: Proposal helmet without mittens and booties
  cooling helmet
Period: Overall Study
Arm/Group | Cryoprotection With Mittens and Booties | Standard Cryoprotection
Started | 141 | 139
Completed | 123 | 120
Not Completed | 18 | 19
Not completed — Inclusion criteria not met | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Protocol Violation | 0 | 4
Not completed — Physician Decision | 2 | 4
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 9 | 8
Not completed — Relapse | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat analysis. 6 patients removed from the analysis because no taxotere treatment was performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoprotection With Mittens and Booties | Standard Cryoprotection | Total
Number analyzed (Participants) | 141 | 133 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11) | 54 (12) | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 133 | 274
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Occurrence of Nail Toxicity of Grade 2 of Common Toxicity Criteria for Adverse Effects V4.0 Evaluated at 8 Weeks Post Infusion of Docetaxel.
Time Frame: 8 weeks post infusion of docetaxel
Population: Intention-to-treat analysis. 6 patients removed from the analysis because no taxotere treatment was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoprotection With Mittens and Booties | Standard Cryoprotection
Number analyzed (Participants) | 141 | 133
Participants | 26 | 49
Statistical Analysis 1: Comparison: Cryoprotection With Mittens and Booties vs Standard Cryoprotection; Test type: Superiority; p < 0.001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: All-Cause mortality was assessed until the last visit (i.e. Consultation 12 months after the last course of Docetaxel), on average 16.5 months
Description: All-Cause mortality monitored/assessed. Serious and Other (Not Including Serious) Adverse Events were not assessed for the study.
Arm/Group | Cryoprotection With Mittens and Booties | Standard Cryoprotection
All-Cause Mortality (participants affected / at risk) | 1/141 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT02283983/Prot_SAP_000.pdf